CLINICAL TRIAL: NCT04726930
Title: High Frequency Ultrasound Spring-load Front-and-side Firing Needle Transducer Developments and Pre-clinical Regional Anesthesia Validation Study
Brief Title: Ultrasound Needle Transducer for Regional Anesthesia Validation Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-04-003B
Record Dates: First submitted 2021-01-26; First posted 2021-01-27 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Thorax; Pain, Spine, With Radicular and Visceral Pain; Acute Post-thoracotomy Pain; Pain, Postoperative; Ultrasound Therapy; Complications
Keywords: Intercostal nerve block; Paravertebral block; Ultrasound-guided pain intervention; Thoracic surgery; Breast surgery; Abdominal surgery; Ultrasound-guided peripheral nerve block; Postoperative pain
MeSH Terms: conditions — Pain; Visceral Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Intercostal nerve block with surface ultrasound: Number of participants: 10 Intercostal blocks will be performed under guidance of surface ultrasound. After we reach the injection site, the puncture stylet will be replace by Intra-needle ultrasound transducer (INUS). Collect signal from Intra-needle ultrasound transducer and then inject local anesthetics.
  Code name: ICNB-INUS-check
  Interventions: Procedure: Intercostal nerve blocks
- Paravertebral block with surface ultrasound: Number of participants: 10 Paravertebral blocks will be performed under guidance of surface ultrasound. After we reach the injection site, the puncture stylet will be replace by Intra-needle ultrasound transducer (INUS). Collect signal from Intra-needle ultrasound transducer and then inject local anesthetics.
  Interventions: Procedure: Paravertebral block
- Intercostal nerve block with intra-needle and surface ultrasound: Number of participants: 10 Intercostal blocks will be performed under guidance of intra-needle "and" surface ultrasound. The intra-needle transducer will be placed inside the puncture needle and it will be the primary guidance to reach target injection site. Surface ultrasound will be the secondary image guide for simultaneous comparison. Collect signal from both Intra-needle ultrasound transducer and surface ultrasound, and then inject local anesthetics.
  Code name: ICNB-INUS-guide
  Interventions: Procedure: Intercostal nerve blocks
- Paravertebral nerve block with intra-needle and surface ultrasound: Number of participants: 10 Paravertebral blocks will be performed under guidance of intra-needle "and" surface ultrasound. The intra-needle transducer will be placed inside the puncture needle and it will be the primary guidance to reach target injection site. Surface ultrasound will be the secondary image guide for simultaneous comparison. Collect signal from both Intra-needle ultrasound transducer and surface ultrasound, and then inject local anesthetics.
  Code name: PVB-INUS-guide
  Interventions: Procedure: Paravertebral block

INTERVENTIONS:
Procedure: Intercostal nerve blocks — Intercostal nerve block is a regional anesthetic procedure for peri-operative pain management. It inhibits the action of the ipsilateral sensory and motor branches, and produces analgesic effects at the targeted thoracic level.
  Other Names: ICNB
  Groups: Intercostal nerve block with intra-needle and surface ultrasound; Intercostal nerve block with surface ultrasound
Procedure: Paravertebral block — Paravertebral block is the technique of injecting local anesthetic alongside the thoracic vertebra close to where the spinal nerves emerge from the intervertebral foramen. This produces unilateral, segmental, somatic, and sympathetic nerve blockade, which is effective for anesthesia and in treating acute and chronic pain of unilateral origin from the chest and abdomen
  Other Names: PVB
  Groups: Paravertebral block with surface ultrasound; Paravertebral nerve block with intra-needle and surface ultrasound

SUMMARY:
To validate the efficacy of miniaturized ultrasound needle transducer as the primary guide for thoracic regional anesthesia.

DETAILED DESCRIPTION:
Paravertebral (PVB) and intercostal nerve block (ICNB) are both techniques of injecting local anesthetics for pain management at thoracic and upper abdominal region.

Today, PVB and ICNB are performed under the guidance of surface two dimensional B-mode ultrasound. However, the procedure still carries potential risks for inexperienced operators since the target zone is very close (2-3 mm) to the pleura. In certain patients, such as those with obesity, the steep needle trajectory and poor quality of the anatomic image make the nerve block even more difficult.

Inaccurate identification of the anatomical structures or suboptimal positioning of the needle tip could result in complications and blockade failure.

We designed an intra-needle ultrasound (INUS) system to improve the identification of anatomical structures and needle tip position. The system passed all safety standards including electrical safety test, biocompatibility test, software certification.

This study is to investigate the feasibility and image quality of INUS during ICNB and PVB. The study protocol is approved and under monitoring for safety and compliance from both Institutional Review Board of Taipei Veterans General Hospital and Ministry of Health and Welfare, Taiwan, Republic of China.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for elective thoracic surgery
2. Patients scheduled for elective upper abdominal surgery
3. Patients scheduled for elective breast surgeries.

Exclusion Criteria:

1. Known coagulopathies,
2. Skin lesion or infection at site of nerve block
3. Pregnant women
4. Allergic to local anesthetics
5. Cognitive diseases
6. Unstable hemodynamics
7. Chronic substance abuse (ex. alcohol, hypnotics, opioids)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Taipei Veterans General Hospital for elective thoracic, upper abdominal, or breast surgeries will be invited to join this trial.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Needling time | Needle insertion to needle withdrawal, up to 20 minutes
  Needle insertion to needle withdrawal (minutes)
Nerve block procedure time | Time from ultrasound contact with skin to needle withdrawal, up to 20 minutes
  How long the procedure takes in minutes, starting from ultrasound contact with skin to needle withdrawal
Success rate of blockade | 20 minutes post administration of local anesthetics (by ultrasound or cold sensation) or intraoperative (at the time of video-thoracoscope exploration)
  Successful blockade will be determined by 1.ultrasound evidence of ideal spreading or 2.evidence of fluid accumulation around intercostal nerves or at paravertebral space under thoracoscope, or 3. loss of cold sensation on the chest or abdomen at block level.
Visibility of needle tip and anatomic structure | During block procedure, up to 60 minutes.
  Record the visibility of needle tip, intercostal muscle, superior costotransverse ligament, pleura. Assessed by the inserting anesthetist on a 5 point Likert scale

SECONDARY OUTCOMES:
Inadvertent pleural puncture or pneumothorax | 20 minutes post-procedure or intraoperative (if needle injuries on pleura noted by thoracoscope)
  Calculate the rate of Inadvertent pleural puncture or pneumothorax, defined by image evidence of pleura injuries or pneumothorax by thoracoscope, X-ray, or CT.

CONTACTS AND LOCATIONS:
Overall Officials: FU-WEI SU, MD, Study Chair — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan, R.o.c., Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Sharing individual participant data that underlie the results reported in future publication, after de-identification ( text, tables, figures)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: three months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal and receive the authors consent.